CLINICAL TRIAL: NCT06833385
Title: Comparative Evaluation of Pediatric Patient Comfort, Time, and Preference Between Digital Scans and Rubber Base Impressions. Crossover Study Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yasmine Ahmed Mortada Abd Elfatah (Other)
Responsible Party: Sponsor-Investigator, Yasmine Ahmed Mortada Abd Elfatah, Lecturer in Pediatric Dentistry and Dental Public Health Departme,Faculty of Dentistry, Assiut University, Assiut, Egypt., Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-2025-0002
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Patient With Early Loss of Primary Teeth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoral Scanning First, PVS Impression Second (Experimental)
  Interventions: Diagnostic Test: Intraoral Scanning; Diagnostic Test: PVS Impression
- PVS Impression First, Intraoral Scanning Second (Experimental)
  Interventions: Diagnostic Test: Intraoral Scanning; Diagnostic Test: PVS Impression

INTERVENTIONS:
Diagnostic Test: Intraoral Scanning — Participants will first undergo intraoral scanning using a digital scanner to capture a 3D image of their dental arches. The procedure is non-invasive and requires no impression material. After one week, the same participants will undergo a polyvinyl siloxane (PVS) impression using conventional impression trays and materials
Diagnostic Test: PVS Impression — Participants will first undergo a polyvinyl siloxane (PVS) impression, where an impression tray filled with PVS material is used to capture the shape of their dental arches. After one week, the same participants will undergo intraoral scanning using a digital scanner for a 3D image of their dentition.

SUMMARY:
The comfort of impression methods and the time they require are important because it is known that children are more stressed in their encounter with the dentist than the elderly, and their chairside times are shorter. The comparison of impression methods in terms of comfort, preference, and time has been studied only in young adults or adult patients. thus this study will assess pediatric patient comfort, time, and preference between digital scans and rubber base impressions.

ELIGIBILITY:
Inclusion Criteria:

* cooperative healthy 6-11 years old child

Exclusion Criteria:

* uncooperative with experience with technique

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Patient Preference for Impression Technique | Immediately after the second impression (within the same visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Dentistry, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient confidentiality concerns and ethical considerations. The collected data is specific to the study objectives and not intended for